CLINICAL TRIAL: NCT04488224
Title: Nano-X Image Guidance: CBCT With Gravity-induced Motion
Acronym: Nano-X IG
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: South Eastern Sydney Local Health District (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: Nano-X IG
Record Dates: First submitted 2020-07-16; First posted 2020-07-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-03

CONDITIONS: Cancer
Keywords: Radiation Therapy; Image Guidance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will undergo CBCT imaging during rotation on the Nano-X patient rotation system. For each participant, quality of CBCT images acquired during the rotation session will be compared with quality of CBCT images collected during their standard radiation therapy treatment.
Who Masked: Outcomes Assessor
Masking Description: The Postdoctoral Research Associate will collect and de-identify CBCT images acquired during Nano-X rotation session and during participants' routine treatment. The software used to display the scans will incorporate a random number generator to determine the labeling of images as 'A' or 'B'. Observers assessing image quality for study outcomes will be masked to the source of either image.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving CBCT Image Guidance during treatment (Experimental): On two separate occasions, CBCT images will be acquired while participants are rotated 360° about the horizontal axis on the Nano-X Patient Rotation System. The rotation will take approximately 72 seconds to complete. Psychometrically validated questionnaires will be completed by the participant before and after each Nano-X CBCT session.
  Participants in this arm undergo conventional CBCT for image guidance during standard of care (SOC) radiotherapy treatment. These participants do not require an additional conventional CBCT as the SOC conventional CBCT images are used to benchmark the experimental Nano-X CBCT scans for evaluation of the primary outcome measure.
  Interventions: Device: Nano-X Patient Rotation System; Other: Psychometrically validated questionnaires
- Patients not receiving CBCT Image Guidance during treatment (Experimental): On two separate occasions, CBCT images will be acquired while participants are rotated 360° about the horizontal axis on the Nano-X Patient Rotation System. The rotation will take approximately 72 seconds to complete. Psychometrically validated questionnaires will be completed by the participant before and after each Nano-X CBCT session.
  Participants in this arm do not undergo conventional CBCT for image guidance during standard of care (SOC) radiotherapy treatment. As such these participants will receive an additional conventional CBCT scan on standard equipment which used to benchmark the experimental NAno-X CBCT scans for evaluation of the primary outcome measure.
  Interventions: Device: Nano-X Patient Rotation System; Radiation: Conventional CBCT scan; Other: Psychometrically validated questionnaires

INTERVENTIONS:
Device: Nano-X Patient Rotation System — The Nano-X prototype is a horizontal patient rotation system that immobilises participants while being rotated on the horizontal axis.
  This device will be used to rotate patients horizontally while cone-beam Computed Tomography (CBCT) projections are acquired.
Radiation: Conventional CBCT scan — A conventional cone-beam Computed Tomography (CBCT) scan is acquired on standard radiotherapy machinery.
  Arms: Patients not receiving CBCT Image Guidance during treatment
Other: Psychometrically validated questionnaires — The Claustrophobia Questionnaire (CLQ), Short Form State/Trait Anxiety inventory (STAI) and Fast Motion Sickness (FMS) questionnaires administered. CLQ only once before the first session, STAI and FMS both before and after each Nano-X CBCT session.

SUMMARY:
A pilot stage, device feasibility trial, to investigate the feasibility of acquiring cone beam computed tomography (CBCT) images for image guidance for radiation therapy by maintaining a fixed imaging system and rotating the participant about the horizontal axis using the Nano-X patient rotation system. It is a single-arm, controlled, single-blinded, non-treatment, non-invasive, single-institution trial.

DETAILED DESCRIPTION:
Primary objective:

To investigate the feasibility of volumetric image guidance for the Nano-X patient rotation system (PRS).

Secondary objectives:

1. To develop image reconstruction methods that allow target and normal tissue visualisation at all treatment angles to a clinical cone beam computed tomography (CBCT) standard.
2. To determine the reproducibility and variability in Nano-X CBCT compared to clinical CBCT.
3. To measure the magnitude of gravity-induced anatomical deformation and translation.
4. To develop treatment plan adaptation methods to compensate for gravity-induced target motion based on Nano-X CBCT image reconstruction at varying treatment angles.
5. To quantify the participant experience of horizontal rotation using the Nano-X PRS for volumetric image guidance CBCT acquisition.

The investigators will perform a pilot stage, device feasibility trial, to investigate the feasibility of acquiring CBCT images for image guidance by maintaining a fixed imaging system and rotating the participant about the horizontal axis using the Nano-X PRS. It is a single-arm, controlled, single-blinded, non-treatment, non-invasive, single-institution trial.

Eligible participants will be asked to attend the Nelune Comprehensive Cancer Centre (NCCC) at the Prince of Wales Hospital on two separate occasions to obtain Nano-X CBCT scans. For each scan the participant will be rotated 360° about the horizontal axis which will take approximately 72 seconds to complete.

Participants will be asked to complete validated psychometric questionnaires before and after each Nano-X CBCT. The questionnaire responses will be used to quantify their experiences of anxiety and motion sickness, and report previous experiences of claustrophobia, in order to identify determinants of tolerance level.

The projection data sets from the Nano-X CBCT scans, along with conventional CBCTs obtained for the participants' standard radiotherapy treatment, will be used to investigate the image-related objectives. The two Nano-X CBCT data sets from each participant will be used to compare Nano-X CBCT variability and reproducibility to clinical CBCT acquisition.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients that are receiving radiation therapy that are able to be imaged with the Nano-X PRS with one of the following tumour sites:

   1. in the head/neck region
   2. in the chest/abdomen/pelvic region with fast CBCT used for standard of care image guidance and is aged 60 years or older
   3. in the chest/abdomen/pelvic region not receiving CBCT for standard of care image guidance and is aged 70 years or older
   4. diagnosis of lung cancer with stage II-IV
2. ≥18 years of age
3. ECOG Performance Status 0-2
4. Must be able to communicate fluently in English to:

   i. Receive instructions from operators of the PRS for safety entering and leaving the Patient Rotation System and required conduct during the during the rotation session, and ii. Communicate their level of comfort or distress to operators of the equipment.
5. Signed, written informed consent or approved alternative, non-contact method for informed consent.

Exclusion Criteria:

1. Pregnant women
2. Patients for whom attaining informed consent would not be possible, including mentally impairment
3. Patients with severe vertigo or recent a diagnosis of Benign Paroxysmal Positioning Vertigo.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Cone Beam Computed Tomography (CBCT) images acquired with horizontal patient rotation that are deemed to be of comparable image quality to clinical CBCT or deemed acceptable for radiotherapy image guidance as scored by a panel of experts. | 6 months
  Observers will view the image sets in 3 orthogonal views and grade the image quality considering geometrical accuracy, anatomical visualisation, sharpness of the image, soft tissue contrast, image noise and uniformity and overall clinical usability.
  The imaging method will be deemed technically feasible if >70% of CBCT images acquired with horizontal patient rotation are deemed of clinical quality.

SECONDARY OUTCOMES:
Change in Short Form State/Trait Anxiety inventory (STAI) and Fast Motion Sickness (FMS) questionnaire scores before and after rotation as assessed by the Wilcoxon signed rank test. | 6 months
  Wilcoxon signed rank test used to determine statistically significant differences in anxiety and motion sickness assessed using psychometrically validated surveys completed prior to and post horizontal rotation CBCT scan.
  The STAI questionnaire is used to assess anxiety and is comprised of 6 questions scored 1-4. These are combined for a final score between 6 and 24, where a higher number indicates a greater level of anxiety.
  The FMS questionnaire is used to assess motion sickness. Participants rate their levels of motion sickness on a scale of 0-20 where 0 is no feeling of nausea and 20 is feeling terrible and very sick.

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Keall, PhD, Principal Investigator — ACRF Image X Institute, University of Sydney; Michael Jackson, MD, Principal Investigator — Prince of Wales Hospital; Simon Downes, MASc, Study Chair — Prince of Wales Hospital; Mark Gardner, PhD, Study Chair — ACRF Image X Institute, University of Sydney

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data may be provided to an external (non-university) research data repository, archive or register with the intention that it be made publicly available for other scientific research. Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/board, under a materials transfer agreement with the university.
Time Frame: This data will become available upon completion of the study.

REFERENCES:
- [Derived] Debrot E, Liu P, Gardner M, Heng SM, Chan CH, Corde S, Downes S, Jackson M, Keall P. Nano X Image Guidance in radiation therapy: feasibility study protocol for cone beam computed tomography imaging with gravity-induced motion. Pilot Feasibility Stud. 2023 Jun 13;9(1):95. doi: 10.1186/s40814-023-01340-z. PMID 37312127